CLINICAL TRIAL: NCT01858519
Title: A Point Prevalence Study to Evaluate the Prevalence of Antibodies to Selected Porcine Viruses in Patients With Cystic Fibrosis Who Are Receiving Porcine-Derived Pancreatic Enzyme Replacement Therapy: A Harmonized Protocol Across Sponsors
Brief Title: Prevalence of Antibodies to Selected Porcine Viruses in Patients With Cystic Fibrosis Receiving Porcine-derived Pancreatic Enzyme Replacement Therapy
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Collaborators: Forest Laboratories (Industry); Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: JSPP-12-01
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Cystic Fibrosis
Keywords: pancreatic enzyme replacement therapy; antibodies; porcine viruses; epidemiology; prospective
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum specimens for subsequent assay for antibodies to HEV and other selected porcine viruses
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CF patients receiving PERT: Cystic fibrosis (CF) patients receiving pancreatic enzyme replacement therapy (PERT)
- Matched control patients unexposed to PERT: Patients unexposed to pancreatic enzyme replacement therapy (PERT); matched on age and location of residence to PERT-exposed CF patients with chronic disease.

SUMMARY:
This is a point prevalence study conducted entirely in the United States (US) to establish the prevalence of antibodies to hepatitis E virus (HEV) and other selected porcine viruses in cystic fibrosis (CF) patients receiving pancreatic enzyme replacement therapy (PERT) for pancreatic insufficiency compared with matched (age and region of residence) control patients with chronic medical conditions unexposed to PERT.

DETAILED DESCRIPTION:
This is a multicenter, non-interventional point-prevalence study conducted in the US to determine the seroprevalence of antibodies to selected porcine viruses in pancreatic enzyme replacement therapy-exposed CF patients and in an unexposed control group with chronic medical conditions matched for age and geographic region of residence. Data collection includes demographic and medical history, pancreatic enzyme replacement therapy, transfusion history, and history of potential exposure to pig viruses. If a patient meets all the requirements of the study and provides a study specific informed consent/assent, a single blood sample is obtained as part of a planned standard-of-care blood collection.

This harmonized protocol reflects equal sponsorship not only by the registering Sponsor, AbbVie, but also the Collaborators, Aptalis Pharma and Janssen Research & Development, LLC.

ELIGIBILITY:
Inclusion Criteria:

All Patients (PERT-exposed and unexposed controls) must meet the following criteria:

* Have a blood draw planned as part of their standard of care following enrollment into the study; and
* Provide informed consent/assent.

Patients in the PERT-Exposed Group must meet the following criteria:

* Have been diagnosed with CF; and
* Have received PERT for a minimum of 6 months.

Patients in the Unexposed Control Group must meet the following criteria:

* Be under medical management for chronic disease;
* Never received any PERT product; and
* Match an enrolled PERT-exposed patient based on age and region-of-residence.
* Have a blood draw planned to be performed within 180 days of the matched PERT-exposed patient blood draw.

Exclusion Criteria:

* Has a porcine heart valve, a porcine-derived graft, or has had exposure to porcine derived insulin. This exclusion does not apply to previous porcine-derived heparin exposure. ;
* Refuses blood collection; or
* Has any condition that, in the opinion of the investigator, would make participation not be in the best interest (e.g., compromise the well-being) of the patient or that could prevent, limit, or confound the protocol-specified assessments.

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cystic fibrosis (CF) patients receiving pancreatic enzyme replacement therapy (PERT) and patients with chronic disease not receiving any PERT.
Sampling Method: Non-Probability Sample
Enrollment: 1310 (Actual)
Dates: Start 2013-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Seroprevalence of antibodies to hepatitis E virus (HEV) and other selected porcine viruses | 18 Months
  Seroprevalence of antibodies to selected porcine viruses in cystic fibrosis (CF) patients exposed to porcine-derived pancreatic enzyme replacement therapy (PERT) compared with a 1:1 matched control group of patients with chronic disease unexposed to PERT

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard J Leitz, MD, Study Director — Janssen Research & Development, LLC
Locations (47):
- United States (47):
  - Site Reference ID/Investigator# 116382, Anchorage, Alaska
  - Site Reference ID/Investigator# 116444, Little Rock, Arkansas
  - Site Reference ID/Investigator# 116595, Long Beach, California
  - Site Reference ID/Investigator# 116855, Los Angeles, California
  - Site Reference ID/Investigator# 116879, Los Angeles, California
  - Site Reference ID/Investigator# 116448, Los Angeles, California
  - Site Reference ID/Investigator# 154681, Denver, Colorado
  - Site Reference ID/Investigator# 116441, Hartford, Connecticut
  - Site Reference ID/Investigator# 127584, New Haven, Connecticut
  - Site Reference ID/Investigator# 116440, Gainesville, Florida
  - Site Reference ID/Investigator# 116882, Miami, Florida
  - Site Reference ID/Investigator# 116277, Orlando, Florida
  - Site Reference ID/Investigator# 116435, Tampa, Florida
  - Site Reference ID/Investigator# 131935, Atlanta, Georgia
  - Site Reference ID/Investigator# 116452, Boise, Idaho
  - Site Reference ID/Investigator# 116442, Chicago, Illinois
  - Site Reference ID/Investigator# 116465, Maywood, Illinois
  - Site Reference ID/Investigator# 141881, Niles, Illinois
  - Site Reference ID/Investigator# 127295, Peoria, Illinois
  - Site Reference ID/Investigator# 116877, Indianapolis, Indiana
  - Site Reference ID/Investigator# 116436, Wichita, Kansas
  - Site Reference ID/Investigator# 136816, Louisville, Kentucky
  - Site Reference ID/Investigator# 116450, New Orleans, Louisiana
  - Site Reference ID/Investigator# 116455, Shreveport, Louisiana
  - Site Reference ID/Investigator# 116461, Boston, Massachusetts
  - Site Reference ID/Investigator# 116463, Grand Rapids, Michigan
  - Site Reference ID/Investigator# 116445, Jackson, Mississippi
  - Site Reference ID/Investigator# 116883, Omaha, Nebraska
  - Site Reference ID/Investigator# 116876, Buffalo, New York
  - Site Reference ID/Investigator# 130461, New Hyde Park, New York
  - Site Reference ID/Investigator# 116449, Syracuse, New York
  - Site Reference ID/Investigator# 116458, Cincinnati, Ohio
  - Site Reference ID/Investigator# 116276, Toledo, Ohio
  - Site Reference ID/Investigator# 116464, Oklahoma City, Oklahoma
  - Site Reference ID/Investigator# 116457, Hershey, Pennsylvania
  - Site Reference ID/Investigator# 116880, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 116467, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 116466, Pittsburgh, Pennsylvania
  - Site Reference ID/Investigator# 116462, Charleston, South Carolina
  - Site Reference ID/Investigator# 116453, Sioux Falls, South Dakota
  - Site Reference ID/Investigator# 116875, Knoxville, Tennessee
  - Site Reference ID/Investigator# 116856, Houston, Texas
  - Site Reference ID/Investigator# 116459, Tyler, Texas
  - Site Reference ID/Investigator# 116278, Norfolk, Virginia
  - Site Reference ID/Investigator# 116460, Richmond, Virginia
  - Site Reference ID/Investigator# 116438, Morgantown, West Virginia
  - Site Reference ID/Investigator# 116439, Madison, Wisconsin

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/pancrelipase_JSPP-12-01.pdf